CLINICAL TRIAL: NCT06910228
Title: Changes in Cerebral Oxygenation Related to Intraoperative Position Changes
Status: Enrolling by invitation | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief - Department of Anesthesiology and Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00004900
Record Dates: First submitted 2025-04-02; First posted 2025-04-04 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Scoliosis Patients
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Near infrared spectroscopy (NIRS) — A non-invasive technique that uses light to assess brain function and tissue oxygenation.

SUMMARY:
This is a prospective, observational study. This study will assess the effect of temporary changes in body position (supine, head of bed elevated 30 degrees, head of bed elevated 60 degrees) in anesthetized patients. Tissue oxygenation will be assessed non-invasively using near infrared spectroscopy (NIRS) by a device that is used in our operating rooms and the ICU setting to assess cerebral and tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Patients 10-21 years of age undergoing posterior spinal fusion, requiring neurophysiologic monitoring and an arterial cannula

Exclusion Criteria:

* Patients in whom an arterial cannula is not indicated for the surgical procedure
* Patients with comorbid conditions that may impact cerebral blood flow, cerebral perfusion or place them at risk for cerebral hypoperfusion
* Patients in whom an invasive arterial cannula cannot be placed

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients having surgery at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral oxygenation at 30 degrees | 5-10 minutes after start of study
  Moving the head of the bed to 30 degrees and comparing cerebral oxygen levels to levels when patient was lying flat.
Change in cerebral oxygenation at 60 degrees | 10-15 minutes after start of study
  Moving the head of the bed to 60 degrees and comparing cerebral oxygen levels to levels when patient was lying flat.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No